CLINICAL TRIAL: NCT07361146
Title: A Comparative Study of Intradialytic Versus Pre-Dialysis Physical Therapy Interventions in Individuals Undergoing Hemodialysis: A Randomized Controlled Trial
Brief Title: A Comparative Study of Intradialytic vs. Pre-Dialysis Physical Therapy Interventions in Individuals Undergoing Hemodialysis: A Randomized Controlled Trial
Acronym: DIAL-PT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Arian (Other Government)
Responsible Party: Sponsor-Investigator, Mohammad Arian, Principal Investigator, Ministry of Health, Kuwait
Organization: Ministry of Health, Kuwait (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/2681; IRB-2024-2681 (Other: MOH Ethics Committee Approval Number)
Record Dates: First submitted 2026-01-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: End-stage Renal Disease (ESRD); Chronic Kidney Disease; Hemodialysis Patients; Physical Rehabilitation During Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradialytic Physical Therapy (During Dialysis) (Experimental): Participants in this group will perform supervised physical therapy exercises during dialysis sessions twice weekly for 12 weeks (approximately 30 minutes each session, including warm-up, resistance training, and cool-down).
  Interventions: Behavioral: Physical Therapy Exercise Program
- Pre-Dialysis Physical Therapy (Before Dialysis) (Active Comparator): Participants in this group will perform supervised physical therapy exercises before dialysis sessions twice weekly for 12 weeks, following the same exercise protocol and duration as the intradialytic group.
  Interventions: Behavioral: Physical Therapy Exercise Program

INTERVENTIONS:
Behavioral: Physical Therapy Exercise Program — A structured physical therapy program including warm-up, strengthening, balance, and stretching exercises delivered either during or before hemodialysis sessions (twice weekly for 12 weeks).

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of two different timings of physical therapy for individuals undergoing hemodialysis: intradialytic (during dialysis) and pre-dialysis (before dialysis). The study seeks to determine which approach provides better improvements in physical function, quality of life, and biochemical outcomes such as hemoglobin and electrolyte levels.

A total of 72 adult participants with end-stage renal disease (ESRD) receiving hemodialysis will be randomly assigned to one of two groups. Both groups will receive standardized educational sessions on the benefits and safety of exercise before beginning the intervention. Participants in the intradialytic group will perform supervised exercises during their dialysis sessions, while those in the pre-dialysis group will complete similar exercises before their dialysis sessions. Each participant will undergo the intervention twice per week for 12 weeks.

Primary outcomes include physical function, assessed using the Six-Minute Walk Test and the Five Times Sit-to-Stand Test. Secondary outcomes include hemoglobin levels, electrolyte balance, and health-related quality of life measured by the KDQOL questionnaire. The study will be conducted at Mubarak Al-Abdullah Al-Jaber Al-Sabah Dialysis Center, Kuwait, following ethical approval from the Ministry of Health Research Ethics Committee.

The results are expected to inform best practices for integrating physical therapy into dialysis care to enhance the health, safety, and well-being of individuals undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 21 and 65 years.
* Diagnosed with end-stage renal disease (ESRD).
* Undergoing maintenance hemodialysis for at least 3 months.
* Medically stable and cleared by the nephrologist to participate in moderate physical exercise.
* Able to understand and follow verbal instructions and provide informed consent.

Exclusion Criteria:

* Uncontrolled hypertension, recent myocardial infarction, or unstable angina.
* Severe musculoskeletal, neurological, or cardiovascular disorders that limit physical activity.
* Active infection, fever, or open wounds.
* Recent hospitalization within the past month.
* Participation in any other structured exercise program within the last 3 months.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-02 (Actual); Primary Completion 2027-03-02 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test (6MWT) | Baseline, every 4 weeks during the 3-month intervention period, and at 6-month follow-up
  Assessment of functional exercise capacity by measuring the total distance walked in six minutes.
Quality of Life (Kidney Disease Quality of Life - KDQOL) | Baseline, every 4 weeks during the 3-month intervention period, and at 6-month follow-up
  Quality of life assessed using the Kidney Disease Quality of Life (KDQOL) questionnaire.
Five Times Sit-to-Stand Test (FTSST) | Baseline, every 4 weeks during the 3-month intervention period, and at 6-month follow-up
  Assessment of lower limb strength and functional mobility by measuring the time required to complete five sit-to-stand repetitions.

SECONDARY OUTCOMES:
Hemoglobin Level | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Measurement of hemoglobin concentration from blood samples.
Serum Potassium Level | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Measurement of serum potassium concentration.
Serum Sodium Level | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Measurement of serum sodium concentration obtained from routine blood samples.
Serum Calcium Level | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Measurement of serum calcium concentration obtained from routine blood samples.
Serum Phosphorus Level | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Measurement of serum phosphorus concentration obtained from routine blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Mubarak Al-Abdullah Al-Jaber Al-Sabah Dialysis Center, Hawalli, Kuwait

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT07361146/Prot_SAP_000.pdf